CLINICAL TRIAL: NCT00299468
Title: Using the Patient Activation Measure (PAM) to Improve Patient Self-Management of Hypertension
Brief Title: The Effect of the Patient Activation Measure on Chronic Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Visiting Nurse Service of New York (Other)
Responsible Party: Linda Gerber, Weill Medical College of Cornell University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 290-00-0013
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2006-05

CONDITIONS: Hypertension
Keywords: hypertension; home care; patient activation; stages-of-change
MeSH Terms: conditions — Hypertension; Patient Participation

INTERVENTIONS:
Behavioral: Patient Activation Measure Intervention Package

SUMMARY:
We will test - in a chronically ill managed long term care population - the effectiveness of an intervention that provides nurse Care Managers with an inventory of evidence-based practices tailored to patients with different levels of knowledge, skills and confidence to engage in self-care management. Specifically, we will develop a "change package" of evidence-based hypertension (HTN) management strategies geared to patients scoring at the four different stages of activation on the Patient Activation Measure (PAM). We will randomly assign a group of interdisciplinary teams in the managed long-term care plan to intervention or control status and will train the Care Managers on the Intervention teams to use the change package in conjunction with a patient's PAM score to design - with the involvement of the patient - an individualized HTN management plan. We then will assess the impact of the intervention on patient activation and outcomes.

DETAILED DESCRIPTION:
The three main aims of the project are to:

1. Determine whether the PAM-driven intervention increases patients' knowledge and self-management skills, measured by both generic PAM scores and HTN-specific measures developed by the research team.
2. Determine whether the PAM-driven intervention improves HTN patients' systolic and diastolic blood pressure (BP), measured in three ways:

   * Average percent reduction in systolic and diastolic BP.
   * Percent of patients who achieve BP control (defined as <140 systolic and <90 diastolic BP or <130 systolic and <80 diastolic for patients with diabetes or renal disease).
   * Percent of patients with controlled HTN who maintain control.
3. Conduct an analysis to examine implementation of the intervention by trainers and Care Managers in the Intervention group and to understand the barriers and facilitators affecting the implementation process.

   In addition, we will conduct a feasibility study with a subset of Care Managers to determine how the Visual Scan Assessment of Patient Activation might be incorporated into routine assessment and care planning procedures. Therefore, the fourth aim of the project is to:
4. Assess the feasibility and perceived usefulness of the Visual Scan Assessment as a tool to increase feedback to Care Managers on how well they are supporting patient self-care management.

ELIGIBILITY:
Inclusion Criteria:

* active VNS CHOICE patient on one of the 22 Intervention or Control teams at the start of the intervention period,
* in care for less than or equal to 730 days,
* a formal diagnosis of HTN (using appropriate ICD codes recorded in the patient record), and
* English speaking.

Exclusion Criteria:

* moderate or severe cognitive impairment as measured by a six-item short portable mental status assessment
* organic brain disease dx in as one of the top 5 dx as measured by information in OASIS, the uniform home care assessment instrument mandated by the Centers for Medicare and Medicaid Services
* End Stage Renal disease dx as one of the top 5 dx as measured by information in OASIS

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2006-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
changes in patients' PAM scores | six months
differences in patients' HTN knowledge | six months
adherence to HTN medication and diet recommendations | six months
average changes in patients' systolic and diastolic BP | six months
percent of patients who maintain BP control, among those with controlled baseline BP | six months

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Gerber, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Visiting Nurse Service of New York Center for Home Care Policy & Research, New York, New York, United States

REFERENCES:
- See also: Visiting Nurse Service of New York — http://www.vnsny.org
- See also: Weill Medical College of Cornell University — http://www.med.cornell.edu/